CLINICAL TRIAL: NCT03904082
Title: Evaluation of the Efficiency of Erector Spina Plane Block and Serratus Anterior Plane Block for Postoperative Thorasic Pain
Brief Title: Comparison of Postoperative Analgesic Consumption of the Erector Spina Plane Block and Serratus Anterior Plane Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ayse Ulgey, Associated professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019/175
Record Dates: First submitted 2019-03-23; First posted 2019-04-04 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Thoracic Diseases
Keywords: dispne, pain
MeSH Terms: conditions — Thoracic Diseases; Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Erector spinae plane block group (ESP) (Active Comparator): Single- shot ultrasound (Esaote Mylab30) guided ESP block with 15 ml 0.25% bupivacain (Marcain 0.5%, Astra Zeneca, Turkey) at the T4 vertebral level will performed preoperatively to patients in the ESP group (Group I).
  Interventions: Procedure: Erector Spinae Plane block ( Group ı)
- Serratus Anterior Plane Block Group (SAP) (Active Comparator): Single- shot ultrasound (Esaote Mylab30 )guided SAP block with 15 ml 0.25% bupivacain (Marcain 0.5%, Astra Zeneca, Turkey) the T4 vertebral level will performed preoperatively to patients in the SAP group( Group II).
  Interventions: Procedure: Serratus Anterior Plane block ( Group ıı)
- Control Group (Placebo Comparator): The Control group receive no intervetion ( Group III).
  Interventions: Procedure: Control Group (GROUPIII)

INTERVENTIONS:
Procedure: Erector Spinae Plane block ( Group ı) — ESP Block will perform preoperative to all patients in ESP block group. Patients in all groups will provide with intravenous patient- controlled analgesia device containing morphine for postoperative analgesia.
  Arms: Erector spinae plane block group (ESP)
Procedure: Serratus Anterior Plane block ( Group ıı) — SAP Block will perform preoperative to all patients in SAP block group. Patients in all groups will provide with intravenous patient- controlled analgesia device containing morphine for postoperative analgesia.
  Arms: Serratus Anterior Plane Block Group (SAP)
Procedure: Control Group (GROUPIII) — Control group will receive no intervetion. Patients in all groups will provide with intravenous patient- controlled analgesia device containing morphine for postoperative analgesia.
  Arms: Control Group

SUMMARY:
To evaluate the ability of Erector spina Plane block and Serratus Anterior Plane block to decrease postoperative pain and analgesia requirements in patients undergoing thoracotomy.

DETAILED DESCRIPTION:
Thoracic wall nerve blocks such as Erector spina Plane block and Serratus Anterior Plane block have become popular for preoperative pain control in patients undergoing thoracotomy.

ELIGIBILITY:
Inclusion Criteria:

ASA I- ASA II Patients

Exclusion Criteria:

* history of allergy to the study medication
* refusal to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
opioid consumption | 48 hours after surgery
  In the recovery room, all patients will given a patient- controlled analgesia device containing morphine 0.5 mg/ml, set to deliver a 1mg bolus dose of morphine with an 15 min lockout time and 6 mg 1 h limit.Total morphine consumption during the 48 hours postoperative period will recorded at 6 time intervals ( 2, 4, 6, 12, 24, 48. hours).
Verbal analog Pain Scores on rest and movement | 48 hours after surgery
  A Research assistant, blinded to the group allocation, interviewed patients and collected data at 6 time intervals ( 2, 4, 6, 12, 24, 48. hours) in the 48 hours postoperatively. Patients were asked to rate their pain using verbal analog scale, where 0= no pain and 10= worst pain possible.

SECONDARY OUTCOMES:
Incidences of adverse effects (like nausea and vomitting) | 48 hours after surgery
  Incidences of nausea and vomitting during the 48 hours postoperative period will recorded at 6 time intervals (2,4,6,12,24,48. hours)

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Ülgey, MD, Study Director — TC Erciyes University
Locations (1):
- Ayşe Ülgey, Kayseri, Talas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identifed individual participant data for all primary and secondary outcome measures will be made aailable.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be aailable within 10 months of study completion.
Access Criteria: Data accep requests will be rewiewed by an external independent Review Panel.Requesters will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Gurkan Y, Aksu C, Kus A, Yorukoglu UH, Kilic CT. Ultrasound guided erector spinae plane block reduces postoperative opioid consumption following breast surgery: A randomized controlled study. J Clin Anesth. 2018 Nov;50:65-68. doi: 10.1016/j.jclinane.2018.06.033. Epub 2018 Jul 2. PMID 29980005
- [Background] Chin KJ, Adhikary S, Sarwani N, Forero M. The analgesic efficacy of pre-operative bilateral erector spinae plane (ESP) blocks in patients having ventral hernia repair. Anaesthesia. 2017 Apr;72(4):452-460. doi: 10.1111/anae.13814. Epub 2017 Feb 11. PMID 28188621
- [Background] Tulgar S, Senturk O. Ultrasound guided Erector Spinae Plane block at L-4 transverse process level provides effective postoperative analgesia for total hip arthroplasty. J Clin Anesth. 2018 Feb;44:68. doi: 10.1016/j.jclinane.2017.11.006. Epub 2017 Nov 14. No abstract available. PMID 29149734
- Available data/document: Clinical Study Report — http://doi.org/10.1016/j.jclinane.2018.06.033